CLINICAL TRIAL: NCT03848351
Title: The Impact of Correct and Efficient Oral Hygiene Maneuvers on Markers of Systemic Inflammation and Overall Well-being.
Brief Title: Oral Hygiene and Systemic Inflammation (Perio-Hygiene 1.0)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Filippo Graziani, DDS MClinDent PhD, Full Professor of Dentistry, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 984/2019
Record Dates: First submitted 2019-02-15; First posted 2019-02-20 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Intervention Model Description: Single-centre randomized, parallel design, clinical trial with a 1-month follow-up
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessor will not be present during explanation of oral hygiene maneuvers. Moreover, participants will be asked not to mention about techniques and group participation to the outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): 70 patients not receiving oral hygiene instructions or devices and continuing with their routine oral hygiene habits
- Test Group (Active Comparator): 70 patients receiving intense oral hygiene instructions assisted by specific software or devices as well as oral hygiene (OH) tools (electric toothbrush, interdental floss, toothpaste) Thus, interventions will consist of.
  * Oral Hygiene Instruction (OHI)
  * Professional supragingival scaling and polishing
  Interventions: Behavioral: Oral Hygiene Instruction (OHI); Procedure: Professional supragingival scaling and polishing

INTERVENTIONS:
Behavioral: Oral Hygiene Instruction (OHI) — OHI will be given focusing on electric toothbrushing as first instance and subsequently focusing on interdental cleaning. OHI will be delivered by trained dental hygienist/periodontist. In the first phase the clinician will explain and show the technique to the patient. The patient will be then invited to perform the technique. Each phase will be assisted and monitored by the clinician. Overall, this sequence may be repeated as many times as the clinician would deem appropriate.
  Arms: Test Group
Procedure: Professional supragingival scaling and polishing — Patients will receive a session of professional supragingival scaling and polishing, that consists of removal of dental plaque and dental calculus from the surface of a tooth, with great care in performing exclusively coronal maneuver. No instrumentation or exploring of the gingival crevice/ sulcus will be performed. Instrumentation will be performed by a trained dental hygienist/periodontist.
  Arms: Test Group

SUMMARY:
The purpose of the study is to evaluate the impact of oral hygiene changes (drastic plaque and gingival inflammation reduction) on markers of systemic inflammation and indicators of oral health related quality of life and other aspects related to overall well-being.

The primary objective is to assess a possible reduction of systemic inflammation as measured through blood bio-markers one month after drastic changes of plaque accumulation. As primary outcome measure, the level of high-sensitive C-reactive protein (hs-CRP) will be assessed.

DETAILED DESCRIPTION:
This study is a single-center, 2 arms, randomized parallel group double-blind clinical trial with one month follow-up, involving patients with no conditions capable of alteration of the systemic inflammatory levels as measured by C-reactive protein (CRP).

Screening will be actuated through a two-step procedure: a careful dental and medical examination will be collected. Subjects with negative history for the conditions tested will undergo blood testing to further confirm the anamnestic findings. Center investigators will document in a screening log reasons for ineligibility or exclusion of subjects. Thus, subjects fulfilling the inclusion criteria will be invited to participate. Clinical center will enroll probands, assigning a unique study subject number and allocating an opaque randomization envelope.

Informed consent will be obtained by the center investigator who will describe the objectives of the study, the alternatives and risks associated with study participation as well as the possibility to withdraw at any time without compromise for the treatment. Consent procedures and documentation of consent will be performed at the screening visit in the national language of the patient and in accordance with local best practice and regulations.

Patients included in the study will undergo a thorough clinical examination aiming at collecting all the data desired (oral and systemic parameters, blood sampling and questionnaires fulfilment). After examinations, the opaque envelope with associated the code of the patient will be opened identifying whether the patient enters Test or Control group.

Patients will also receive a session of professional supragingival scaling and polishing: instrumentation will be performed by a trained dental hygienist/periodontist with great care in performing exclusively coronal maneuver. No instrumentation or exploring of the gingival crevice/ sulcus will be performed.

Subjects in the Test group will receive a thorough session of oral hygiene instruction (OHI) and a full oral hygiene kit.

OHI will be given focusing on electric toothbrushing as first instance and subsequently focusing on interdental cleaning. OHI will be delivered by trained dental hygienist/periodontist.

OHI will be given directly on the patient's mouth. In the first phase the clinician will explain and show the technique to the patient. The patient will be then invited to perform the technique. Each phase will be assisted and monitored by the clinician. Overall, this sequence may be repeated as many times as the clinician would deem appropriate.

Subjects in the control group will be invited to attend another examination in 4 weeks (T28)

Every week, included subjects in the Test group will attend session of OHI re-enforcement and plaque control in order to achieve optimal plaque control. Ideally a value below 20% should be aimed as shown already to be consistent with findings from our research group.

Patients of both groups will undergo clinical examinations, questionnaires and blood withdrawal. The clinical examinations will be performed by examiners blind to group allocation. Participants will be asked by the study coordinators not to disclose to the examiners whether they belong to Test or Control group.

Any periodontal treatment, or professional scaling will be forbidden after the inclusion (T0). For patient allocated in the Test group any pharmacological treatment prescription, or any devices administration different from this study protocol guidelines will be prohibited. In particular, if the patients, in both test or control group, will have to undergo treatment capable of influencing CRP (statins) this will be highlighted and the patient excluded from the study. If withdrawal for prohibited intervention occurs, a new patient enrolment will be activated.

Individuals will be free to quit the study at any time. Patients who will fail to comply with T28 VISIT will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* male or female, 18 to 79 of age, of any race/ethnicity;
* presence of at least 20 teeth;
* ≤ 2 untreated dental caries;
* presence of relevant plaque accumulation as shown by Full Mouth Plaque Scores (FMBS) >50%.
* presence of relevant periodontal/gingival inflammation as shown by FMBS > 35%

Exclusion Criteria:

* • pregnancy and breast feeding;

  * patients undergoing pharmacological treatment capable of reducing CRP such as statins or chronic anti-inflammatory treatment,
  * current or past (≤ 30 days) systemic or local antibiotic therapy;
  * heavy smokers (over 20 cigarettes per day or pipe or cigar);
  * patients undergoing orthodontic treatment;
  * patients not capable to comply with given instruction or administrative issues related to the study
  * dental or periodontal conditions (e.g., deep caries, periodontal abscess) requiring urgent treatment

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline of High sensitivity C-Reactive Protein (hsCRP) at 1 month | Difference of values of the markers collected at Baseline and 1 month after treatment
  analyzed though blood sampling. Unit of measure: mg/L

SECONDARY OUTCOMES:
Change from baseline of Interleukin 6 at 1 month | Difference of values of the markers collected at Baseline and 1 month after treatment
  analyzed though blood sampling. Unit of measure: nmol/L (ng/mL)
Vitamin D | Collected at Baseline
  analyzed though blood sampling. Unit of measure: nmol/L
Full-mouth plaque score (FMPS) | Measured at Baseline and 1 month after treatment
  Changes in Full-mouth plaque score, measuring the amount of dental plaque on the teeth orally through clinical examination. Unit of measure %. The scale ranges from 0% (minimum value, i.e. plaque absent) to 100% (maximum value: all areas are occupied by plaque). 0% would the ideal value. No sub-scales are included.
Full-mouth bleeding score (FMBS) | Measured at Baseline and 1 month after treatment
  Changes of Full-mouth bleeding score, measuring the number of gingival areas that bleed after gingival probe passage. It is measured orally through clinical examination. Unit of measure %. The scale ranges from 0% (minimum value, i.e. gingival inflammation is absent) to 100% (maximum value: all gingival areas are inflamed). 0% would the ideal value. No sub-scales are included.
Pocket probing depth (PPD) | Measured at Baseline and 1 month after treatment
  Changes in PPD, measured orally through clinical examination. Unit of measure: mm (PPD=distance between the gingival margin and the deepest part of the gingival pocket)
Recession of the gingival margin (REC) | Measured at Baseline and 1 month after treatment
  Changes in REC, measured orally through clinical examination. Unit of measure: mm (REC=distance in mm from the cement-enamel junction (CEJ) to the gingival margin )
Clinical attachment level (CAL) | Measured at Baseline and 1 month after treatment
  Changes in CAL, measured orally through clinical examination. Unit of measure: mm (CAL)
  : calculated as the sum of PPD and REC)
Changes of sum of Oral Health Index Profile-14 | Measured at Baseline and 1 month after trea
  Changes in Oral Health Index Profile-14 measured through administration of specific questionnaire. Each of the 14 questions can be answered with a Likert scale reporting from "never" to "always" translated to 1 and 5 respectively. Thus, a maximum value (sum) of 70.
Changes of sum of Pittsburgh sleep quality index (PSQI) | Measured at Baseline and 1 month after trea
  Changes in PSQI measured through administration of specific questionnaires. It is a validated questionnaire of 19 self-questions aiming at assessing statements grouped in 7 component scores: sleep quality, latency, duration, habitual sleep efficiency, disturbances, uses of sleep medications and day time dysfunction. Component scores range between 0 and 3, with 0= "no difficulty" and 3= "severe difficulty". Total score ranges between 0-21. If the patient has a bed partner it is possible to add 5 questions to be filled by the partner, about the sleep quality of the patient.
Changes of sum of Memory Assessment Clinics - Questionnaire (MAC-Q) | Measured at Baseline and 1 month after treatment
  Changes in MAC-Q measured through administration of specific questionnaire. It is a validated questionnaire of 6 self-questions aiming at assessing the quality of the memory in comparison to the period of high school or college. Each question is rated with a 5-point scale, with 1= "much better now" and 5= "much poorer now". The final question is a global evaluation of the memory, so it has more weight in the scoring system and is evaluated in a 10-point scale. Total score range is comprised between 7 and 35.
Changes of sum of Oxford Happiness Questionnaire (OHQ) | Measured at Baseline and 1 month after treatment
  Changes in 0HQ measured through administration of specific questionnaire. It is a validated questionnaire that includes items presented as a single statement which can be endorsed on a uniform 6-point Likert scale.
Food Frequency Questionnaire (FFQ) | Measured at Baseline and 1 month after treatment
  FFQ measured through administration of specific questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Peric M, Marhl U, Gennai S, Marruganti C, Graziani F. Treatment of gingivitis is associated with reduction of systemic inflammation and improvement of oral health-related quality of life: A randomized clinical trial. J Clin Periodontol. 2022 Sep;49(9):899-910. doi: 10.1111/jcpe.13690. Epub 2022 Jul 17. PMID 35762095